CLINICAL TRIAL: NCT00877968
Title: Glycemic Responses and Sensory Characteristics of Whole Yellow Pea Flour Added to Novel Functional Foods
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Pulse Canada (Other)
Responsible Party: Dr. Peter J.H. Jones Professor, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B2008:017
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes
Keywords: Pea flour; Glycemic response; Diabetes; Sensory; Functional food; Diabetes control and prevention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Whole wheat banana bread (Placebo Comparator): Banana bread made with whole wheat flour
  Interventions: Dietary Supplement: Whole wheat banana bread
- Whole pea flour banana bread (Active Comparator): Banana bread made with whole pea flour
  Interventions: Dietary Supplement: Whole pea flour banana bread
- Whole wheat biscotti (Placebo Comparator): Biscotti made with whole wheat flour
  Interventions: Dietary Supplement: Whole wheat biscotti
- Whole pea biscotti (Active Comparator): Biscotti made with whole pea flour
  Interventions: Dietary Supplement: Whole pea flour biscotti
- Whole wheat pasta (Placebo Comparator): Pasta made with whole wheat durum
  Interventions: Dietary Supplement: Whole wheat pasta
- Whole pea flour (Active Comparator): Pasta made with 30% whole pea flour and 70% white wheat durum
  Interventions: Dietary Supplement: Whole pea pasta
- White bread (Placebo Comparator)
  Interventions: Dietary Supplement: White bread
- Boiled yellow peas (Placebo Comparator)
  Interventions: Dietary Supplement: Boiled yellow peas

INTERVENTIONS:
Dietary Supplement: Whole wheat banana bread — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 62.8 g Available CHO: 51.7 g
  Arms: Whole wheat banana bread
Dietary Supplement: Whole pea flour banana bread — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 67.8 g Available CHO: 52.0 g
  Arms: Whole pea flour banana bread
Dietary Supplement: Whole wheat biscotti — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 79.8 g Available CHO: 53.1 g
  Arms: Whole wheat biscotti
Dietary Supplement: Whole pea flour biscotti — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 86 g Available CHO: 51.7 g
  Arms: Whole pea biscotti
Dietary Supplement: Whole wheat pasta — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion (Dry): 70 g Available CHO: 51.1 g
  Arms: Whole wheat pasta
Dietary Supplement: Whole pea pasta — Dose was portioned so that subjects received 50 g available carbohydrate Pea pasta is 30% whole pea pasta, 70 white wheat durum
  Portion (Dry pasta) : 90 g Available CHO: 53.1 g
  Arms: Whole pea flour
Dietary Supplement: White bread — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 100 g Available CHO: 50 g
  Arms: White bread
Dietary Supplement: Boiled yellow peas — Dose was portioned so that subjects received 50 g available carbohydrate
  Portion: 100 g (dry) --> 250 g cooked Available CHO: 52.8 g
  Arms: Boiled yellow peas

SUMMARY:
The objective of this study was to determine if whole yellow pea flour reduces post-prandial glycemic responses of novel food products. The second objective was to determine if whole yellow pea flour produces food products with favorable sensory characteristics including appearance, taste, smell, texture and overall acceptability, compared to corresponding food products made with whole wheat flour.

DETAILED DESCRIPTION:
Pulses, including yellow peas, are readily available and low-cost commodities that are gaining considerable momentum as functional ingredients possessing health benefits, as these food materials are high in fiber, protein, antioxidants, and low in fat. As incidence rates of type II diabetes continue to climb, new novel ingredients that produce low-glycemic food products are in demand. Consumption of whole pulses have been shown to lower post-prandial glycemic responses (Jenkins and others 1983), however, their addition to foods often produces unfavorable sensory characteristics. To date, few studies have examined the feasibility of producing food products containing pulse-derived ingredients that reduce post-prandial glycemic responses, lower glycemic indexes (GI) and at the same time possess sensory qualities that appeal to consumers. Since yellow peas are readily available and relatively inexpensive, they are a promising candidate for use as novel ingredients for the development of low-glycemic, consumer-friendly functional foods.

The objective of the present study was to first determine the post-prandial glycemic response and GI of novel foods containing whole yellow pea flour (WYPF) as a functional ingredient. The second objective was to determine the acceptability of sensory characteristics for each WYPF food product.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* non-lactating women
* BMI's between 18 and 31 kg/m2

Exclusion Criteria:

* heart disease
* diabetes
* thyroid disease
* celiac disease
* gluten intolerance
* taking corticosteroid medications
* smokers
* Chronic alcohol usage (> 2 drinks/d)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemic response

SECONDARY OUTCOMES:
Comparison of hedonic sensory characteristics between corresponding food products
Appearance, taste, texture, smell and overall acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Marinangeli CP, Kassis AN, Jones PJ. Glycemic responses and sensory characteristics of whole yellow pea flour added to novel functional foods. J Food Sci. 2009 Nov-Dec;74(9):S385-9. doi: 10.1111/j.1750-3841.2009.01347.x. PMID 20492127